CLINICAL TRIAL: NCT06175689
Title: Evaluating the Performance of Invasive Ventilation During Specialized Cardiopulmonary Arrest Resuscitation: a Multicentre Observational Study
Brief Title: Evaluating the Performance of Invasive Ventilation During Specialized CPR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: University Hospital, Grenoble (Other); Hôpital Necker-Enfants Malades (Other); Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: CPR CPV
Record Dates: First submitted 2023-10-09; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cardiopulmonary Arrest; Mechanical Ventilation Complication
Keywords: CPR; Cardiopulmonary Arrest; Mechanical ventilation; Volume ventilation; Pressure ventilation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describe the ventilation patterns, describe the evolution of ventilation over time and describe the safety data for two strategies of ventilation (volume or pression modes) during specialized cardiopulmonary resuscitation of pre-hospital cardiorespiratory arrest: an observational and multicentre study.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest is a real public health issue, whose annual incidence in Europe is 67 to 170 per 110,000 inhabitants, but whose survival remains extremely low, of the order of 4.6 to 8%. Rapid implementation of the survival chain and then specialized resuscitation is therefore essential. The recommendations of the 2020 American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care and the 2021 European Rescucitation Council Guidelines recently reaffirmed the quality criteria for cardiopulmonary resuscitation (CPR) basic. Thus, during this CPR, rescuers must perform optimal chest compressions, that is, at a depth of 5 cm without exceeding 6 cm and at a frequency of 100 to 120/min with the minimum interruption time. Decompression must also be of quality.

As regards the ventilation of cardiac arrest, areas of uncertainty persist. This can be done using a bag valve mask (BAVU) or a respirator, regardless of the environment. The oxygen inspired fraction (FiO2) should be as high as possible during CPR. In the case of specialized and medicalized CPR, artificial ventilation must be implemented as soon as possible. Once the orotracheal intubation is performed, the clinician must mechanically ventilate the patient at a frequency of 10 breaths per minute without interrupting chest compressions. A ventilation strategy with reduced tidal volume (6-7 mL.kg-1 weight predicted) is preferred, associated with a low positive tele-expiratory pressure (PEEP) of 0 to 5 cmH20. Despite these clear recommendations, a heterogeneity of ventilatory practices is observed.

Regarding specialized ventilator ventilation, different ventilatory strategies are available for the clinician, however the scientific literature remains poor on this subject, especially in terms of safety and effectiveness of these strategies. Volume-assisted ventilation (VAC) is the most frequently used ventilatory strategy in the world, with the theoretical advantage of controlling the volume delivered to the patient, without being able to guarantee the pressures. Other alternative modes regulated in pressure exist but have the disadvantage of not guaranteeing volumes and minute ventilation. Each of these strategies (volume or pressure mode) is used in common practice, often with a preference for this or that ventilatory technique depending on the center and the available equipment.

The investigators therefore consider it important to accurately assess the ventilatory performance of these two strategies throughout CPR.

To do this, the investigators will conduct an observational, multicentre study. This study will aim to describe the ventilation patterns, describe the evolution of ventilation over time and finally to describe the safety data, for these two strategies during specialized cardiopulmonary resuscitation of pre-hospital cardiorespiratory arrest.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or older)
* With out-of-hospital cardiorespiratory arrest
* For which specialized cardiopulmonary resuscitation is indicated and started
* Supported by the SMUR of the Angers University Hospital of Angers, the Necker-Enfants malades University Hospital, the Grenoble University Hospital and the hospital of Annecy-Genevois
* And for which invasive mechanical ventilation on Monnal T60 transport respirator is started

Exclusion Criteria:

* patients for whom it is decided not to perform invasive ventilation and
* Patients opposed to participating in research
* Patients with a limitation of active therapies
* Patients who are not members or beneficiaries of a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied is that of out-of-hospital cardiorespiratory arrests managed by the emergency medicine prehospital medical teams (SMUR) of the four inclusion centers and meeting the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of minute ventilation depending on capnogram analysis (CO2 patterns) | 12 hours
  Actual minute ventilation (L/min) associated with the predefined CO2 patterns, expressed in L/min/pattern

SECONDARY OUTCOMES:
Description of ventilation | 12 hours
  * active ventilation expressed in percentage of minute ventilation
  * passive ventilation expressed in percentage of minute ventilation
Description of capnogram CO2 patterns | 12 hours
  Distribution of each predefined CO2 patterns expressed in percentage of capnograms recorded per patient.
Description of CPR quality in terms of chest compressions frequency | 12 hours
  Chest compressions frequency analysis will be expressed in time during which chest compression frequency (fCT) is within the predefined ranges (100 to 120 compressions/min) expressed in percentage.
Description of CPR quality in terms of time spent to continuous compressions | 12 hours
  CPR quality criteria analysis will be based in this analysis on CPR fraction (%CT), expressed in percentage, that expresses the percentage of time spent to continuous chest compressions over the total time of cardiopulmonary resuscitation.
Description of initial cardiac rhythm during CPR | 12 hours
  Cardiac rhythm will be expressed in percentage of the entire population
Description of return of spontaneous circulation (ROSC) | 12 hours
  Presence of return of spontaneous circulation (ROSC) will be expressed in percentage of the entire population
Survival at hospital arrival | 12 hours
  Survival at hospital arrival will be expressed in percentage of the entire population
Description of cardiac arrest etiologies characteristics | 12 hours
  Proportion of cardiac arrest etiologies will be expressed in percentages of the entire population
Description of presence of lay-rescuers CPR | 12 hours
  Proportion of presence of lay-rescuers will be expressed in percentages of the entire population
Description of initiation of CPR by-first aid | 12 hours
  Proportion of initiation of CPR first-aid will be expressed in percentages of the entire population
Description of use of automated chest compressions devices | 12 hours
  Proportion of use of automated chest compressions devices will be expressed in percentages of the entire population
Description of use of defibrillators | 12 hours
  Proportion of use of defibrillators will be expressed in percentages of the entire population
Description of use of Extra Corporeal cardio Pulmonary Resuscitation (ECPR) | 12 hours
  Proportion of use of Extra Corporeal cardio Pulmonary Resuscitation (ECPR) will be expressed in percentages of the entire population
Observation of ventilation major events | 12 hours
  Ventilation major events will be defined in percentage of the entire population:
  * Occurence of extubation expressed in percentage
  * Triggering of high pressure alarm expressed in percentage
  * Triggering of low volume (expired volume) alarm expressed in percentage
  * Occurence of hemoptysis in intubation sonde expressed in percentage
  * Occurence of pulmonary edema expressed in percentage

REFERENCES:
- [Background] Perkins GD, Graesner JT, Semeraro F, Olasveengen T, Soar J, Lott C, Van de Voorde P, Madar J, Zideman D, Mentzelopoulos S, Bossaert L, Greif R, Monsieurs K, Svavarsdottir H, Nolan JP; European Resuscitation Council Guideline Collaborators. European Resuscitation Council Guidelines 2021: Executive summary. Resuscitation. 2021 Apr;161:1-60. doi: 10.1016/j.resuscitation.2021.02.003. Epub 2021 Mar 24. PMID 33773824
- [Background] Hubert H, Tazarourte K, Wiel E, Zitouni D, Vilhelm C, Escutnaire J, Cassan P, Gueugniaud PY; GR- ReAC. Rationale, methodology, implementation, and first results of the French out-of-hospital cardiac arrest registry. Prehosp Emerg Care. 2014 Oct-Dec;18(4):511-9. doi: 10.3109/10903127.2014.916024. Epub 2014 May 30. PMID 24877567
- [Background] Merchant RM, Topjian AA, Panchal AR, Cheng A, Aziz K, Berg KM, Lavonas EJ, Magid DJ; Adult Basic and Advanced Life Support, Pediatric Basic and Advanced Life Support, Neonatal Life Support, Resuscitation Education Science, and Systems of Care Writing Groups. Part 1: Executive Summary: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S337-S357. doi: 10.1161/CIR.0000000000000918. Epub 2020 Oct 21. No abstract available. PMID 33081530
- [Background] Considine J, Gazmuri RJ, Perkins GD, Kudenchuk PJ, Olasveengen TM, Vaillancourt C, Nishiyama C, Hatanaka T, Mancini ME, Chung SP, Escalante-Kanashiro R, Morley P. Chest compression components (rate, depth, chest wall recoil and leaning): A scoping review. Resuscitation. 2020 Jan 1;146:188-202. doi: 10.1016/j.resuscitation.2019.08.042. Epub 2019 Sep 16. PMID 31536776
- [Background] Stiell IG, Brown SP, Nichol G, Cheskes S, Vaillancourt C, Callaway CW, Morrison LJ, Christenson J, Aufderheide TP, Davis DP, Free C, Hostler D, Stouffer JA, Idris AH; Resuscitation Outcomes Consortium Investigators. What is the optimal chest compression depth during out-of-hospital cardiac arrest resuscitation of adult patients? Circulation. 2014 Nov 25;130(22):1962-70. doi: 10.1161/CIRCULATIONAHA.114.008671. Epub 2014 Sep 24. PMID 25252721
- [Background] Stiell IG, Brown SP, Christenson J, Cheskes S, Nichol G, Powell J, Bigham B, Morrison LJ, Larsen J, Hess E, Vaillancourt C, Davis DP, Callaway CW; Resuscitation Outcomes Consortium (ROC) Investigators. What is the role of chest compression depth during out-of-hospital cardiac arrest resuscitation? Crit Care Med. 2012 Apr;40(4):1192-8. doi: 10.1097/CCM.0b013e31823bc8bb. PMID 22202708
- [Background] Edelson DP, Abella BS, Kramer-Johansen J, Wik L, Myklebust H, Barry AM, Merchant RM, Hoek TL, Steen PA, Becker LB. Effects of compression depth and pre-shock pauses predict defibrillation failure during cardiac arrest. Resuscitation. 2006 Nov;71(2):137-45. doi: 10.1016/j.resuscitation.2006.04.008. Epub 2006 Sep 18. PMID 16982127
- [Background] Babbs CF, Kemeny AE, Quan W, Freeman G. A new paradigm for human resuscitation research using intelligent devices. Resuscitation. 2008 Jun;77(3):306-15. doi: 10.1016/j.resuscitation.2007.12.018. Epub 2008 Mar 7. PMID 18329159
- [Background] Henlin T, Michalek P, Tyll T, Hinds JD, Dobias M. Oxygenation, ventilation, and airway management in out-of-hospital cardiac arrest: a review. Biomed Res Int. 2014;2014:376871. doi: 10.1155/2014/376871. Epub 2014 Mar 3. PMID 24724081
- [Background] Vissers G, Soar J, Monsieurs KG. Ventilation rate in adults with a tracheal tube during cardiopulmonary resuscitation: A systematic review. Resuscitation. 2017 Oct;119:5-12. doi: 10.1016/j.resuscitation.2017.07.018. Epub 2017 Jul 21. PMID 28739281
- [Background] Cordioli RL, Grieco DL, Charbonney E, Richard JC, Savary D. New physiological insights in ventilation during cardiopulmonary resuscitation. Curr Opin Crit Care. 2019 Feb;25(1):37-44. doi: 10.1097/MCC.0000000000000573. PMID 30531537
- [Background] Cordioli RL, Brochard L, Suppan L, Lyazidi A, Templier F, Khoury A, Delisle S, Savary D, Richard JC. How Ventilation Is Delivered During Cardiopulmonary Resuscitation: An International Survey. Respir Care. 2018 Oct;63(10):1293-1301. doi: 10.4187/respcare.05964. Epub 2018 May 8. PMID 29739857